CLINICAL TRIAL: NCT02957669
Title: Evaluation of Practice Self-Regulation (PS-R)
Brief Title: Evaluation of Practice Self-Regulation
Acronym: PS-R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Policy & Research Group (Other)
Collaborators: The Office of Adolescent Health, HHS (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5 TP1AH000003-02-00 PS-R
Record Dates: First submitted 2016-11-03; First posted 2016-11-08 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Teen Pregnancy Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Practice Self-Regulation (PS-R) (Experimental): Practice Self-Regulation (PS-R) is the treatment condition. PS-R is an in-person, individual-level, clinic-based intervention that aims to increase knowledge of sexual health and the impact of trauma on sexual decision-making.
  Interventions: Behavioral: Practice Self-Regulation
- Therapy Practice Group (Active Comparator): Therapy Practice Group is the control counterfactual condition. It is an individual-level, therapy as usual in which the therapist addresses mental health concerns of the participant.
  Interventions: Behavioral: Therapy Practice Group

INTERVENTIONS:
Behavioral: Practice Self-Regulation — PS-R is an in-person, individual-level, clinic-based intervention implemented by mental health professionals trained in the intervention. It is intended to be implemented in ten structured, individual therapy sessions lasting approximately 50 minutes over the course of 18 weeks.
  Arms: Practice Self-Regulation (PS-R)
Behavioral: Therapy Practice Group — Therapy Practice Group is the control condition aimed at providing the youth a safe space to work on meeting their mental health goals. It is intended to be at least ten sessions over the course of 18 weeks.
  Arms: Therapy Practice Group

SUMMARY:
The purpose of the study is to determine the impact of the offer to participate in the Practice Self-Regulation (PS-R) (treatment) relative to the offer to participate in the Therapy Practice Group (control) on participants' reported number of sexual partners and reported number of times having sex without a condom nine months after the end of treatment.

DETAILED DESCRIPTION:
The Policy & Research Group (PRG) will be evaluating the Practice Self-Regulation (PSR) program. This intervention is designed to address gaps in the existing evidence, reduce disparities in teen pregnancy and associated sexual and reproductive health outcomes, and serve high-need populations. The intervention is composed of ten structured, individual therapy sessions intended to promote optimal sexual decision making. By increasing knowledge of sexual health and the impact of trauma on sexual decision-making, youth are encouraged and supported in practicing self-regulation. The primary focus of the study will be to investigate the impact of the intervention on participants' self-reported sexual behaviors (times having sex with no condom and number of sexual partners). In addition, the study will include exploratory investigations of the following theoretically relevant antecedents to behavior and pathways to behavior change: (1) perception of risk and severity for pregnancy and HIV/STIs; (2) intention to have sex; (3) importance of having sex; (4) intention to use effective contraceptive methods (including condoms); (5) affect regulation self-efficacy; (6) importance of using effective contraceptive methods; (7) intention to limit number of sexual partners; (8) importance to limiting the number of sexual partners; (9) intention to practice affect regulation; (10) self-esteem; (11) importance of using affect regulation; (12) intention to practice sexual self-regulation; (13) importance of practicing sexual self-regulation; (14) contraceptive use and negotiation (including condoms) self-efficacy; (15) sexual activity decision making and planning self-efficacy; (16) beliefs regarding the malleability of emotions; (17) beliefs regarding value of affect regulation; (18) use of effect regulation; and (19) distress . The control (counterfactual) condition, Therapy Practice Group, consists of therapy as usual without the incorporation of elements vital to the PSR intervention. All eligible individuals who provide the proper consent to participate are randomized and enrolled into the study at the time they attend their first scheduled study session. Outcomes will be assessed using self-reported, participant-level data gathered (by way of a questionnaire) at three time points: baseline (enrollment); post-program (immediately after the end of the intervention period, which is 18 weeks after baseline); and 9-month follow-up (9 months following the end of the intervention period, which is 13 months after baseline). The study is taking place in California, Louisiana, New Mexico, Michigan, and Maine. Recruitment of study participants and delivery of the intervention is conducted by trained private practitioners and therapists working at participating agencies who are serving youth between the ages of 14 and 19 and are receiving outpatient mental health services.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 14-19
* Provide parental consent (if under age 18) and participant assent to participate in the study
* Deemed appropriate for the study by the agency staff
* Receiving individual outpatient counseling services at one of the study's implementation sites

Exclusion Criteria:

* Previous participation in the study
* Previous use of the Trauma Outcome Process (TOP) workbook in therapy
* Self-report of previous participation in other TPP-funded programs
* Self-report of roommate who participated in the study

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 432 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
Number of sexual partners | 9 months after the end of the intervention
  Participant self-report of the number of sexual partners in the past three months. Measured through two survey questions which ask the participant with whom they have had sexual contact during their life, and if sexual contact with any gender is reported are subsequently asked how many sexual partners they have had in the past three months.
Times having sex without a condom | 9 months after the end of the intervention
  Participant self-report on the number of times they have had vaginal, oral, or anal sex without a condom in the last three months. Measured through three survey questions which ask the participant how many times they have had vaginal, oral, and anal sex in the past three months.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jenner, PhD, MMC, BA, Principal Investigator — The Policy & Research Group

IPD SHARING:
Plan to Share IPD: Yes
A dataset will be prepared at the conclusion of the study, which includes de-identified individual-level data on all study participants who contributed self-report data. Respondents will be represented only by a research ID number. Included in the dataset will be self-report data collected across all survey administrations (including demographic characteristics, sexual behaviors, and theoretical antecedents to those behaviors) and select information on program participation (e.g., which program sessions were attended). Basic data cleaning steps will be taken in order to ensure data are unidentifiable and to increase usability.
Time Frame: The individual participant dataset will become available twelve months after the study has concluded.

REFERENCES:
- See also: The Policy & Research Group website — http://www.policyandresearch.com/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/69/NCT02957669/Prot_SAP_001.pdf